CLINICAL TRIAL: NCT07224399
Title: A Phase 1, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of BGM1812 Injection Following Single and Multiple Subcutaneous Administration in Normal to Overweight or Obese But Otherwise Healthy Men and Women
Brief Title: Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of BGM1812 Injection Following Single and Multiple Subcutaneous Administration in Normal to Overweight or Obese But Otherwise Healthy Men and Women
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGM1812-P1-CPK01-US
Record Dates: First submitted 2025-10-29; First posted 2025-11-04 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-08

CONDITIONS: Healhty; Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BGM1812 (Part A) (Experimental): Single ascending doses of BGM1812 administered subcutaneously (SC).
  Interventions: Drug: BGM1812
- Placebo (Part A) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo
- BGM1812 (Part B) (Experimental): Multiple ascending doses of BGM1812 administered SC.
  Interventions: Drug: BGM1812
- Placebo (Part B) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGM1812 — Administered SC.
  Arms: BGM1812 (Part A)
Drug: Placebo — Administered SC.
  Arms: Placebo (Part A)
Drug: BGM1812 — Administered SC.
  Arms: BGM1812 (Part B)
Drug: Placebo — Administered SC.
  Arms: Placebo (Part B)

SUMMARY:
This is a Phase 1, single-center, double-blind, placebo-controlled, dose-escalation study. The study will evaluate the pharmacokinetics (PK), pharmacodynamic (PD), preliminary efficacy, safety and tolerability of BGM1812 following single and multiple SC administrations in normal to overweight or obese but otherwise healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the written informed consent document; willingly provides valid, signed written informed consent; willing and able to comply with the schedule, requirements and restrictions of the study.
* Body mass index (BMI) meeting one of the following requirements:

  1. Between ≥ 30.0 kg/m2 and ≤ 40.0 kg/m2 (obese) (for Cohort 3-6); OR
  2. Between ≥ 27.0 kg/m2 and < 30.0 kg/m2 (overweight) with at least 1 of the following: One or more symptoms of prediabetes (impaired fasting plasma glucose and/or abnormal glucose tolerance), grade 1 hypertension, simple fatty liver or dyslipidemia (For Cohort 3- 6); OR
  3. Between ≥ 23.0 kg/m2 and < 27.0 kg/m2 healthy subjects (for Cohort 1 and Cohort 2)
* Have a stable body weight (<5% self-reported change during the previous 12 weeks) before screening

Exclusion Criteria:

* Have allergic predisposition (allergic to 3 or more foods or drugs), or are allergic to amylin agonist-based therapeutic agents or suffer from severe allergic diseases (asthma, urticaria, eczematous dermatitis).
* Known type I/II diabetes.
* Has underwent gastric bariatric surgery in the past, or has had liposuction or fat removal within 1 year before screening, or plan to have bariatric surgery, liposuction or abdominal fat removal during the study period or other surgery that would obviously affect the body weight.
* History of acute or chronic pancreatitis or pancreatic injury.
* Has any other conditions or disorders deemed unsuitable for including in the study, in the opinion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Number of treatment adverse events | Predose up to 6 weeks (Part A) & 9 weeks (Part B)
  The relationship of each adverse event to the investigational product was assessed by the investigator

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of BGM1812 | Predose through week 6 (Part A) & week 9 (Part B)
  PK: AUC of BGM1812
PK: Maximum Observed Concentration (Cmax) of BGM1812 | Predose through week 6 (Part A) & week 9 (Part B)
  PK: Cmax of BGM1812
Pharmacodynamics (PD): Change from baseline in fasting body weight | Predose through week 6 (Part A) & week 9 (Part B)
  Pharmacodynamics (PD): Change from baseline in fasting body weight

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC, Inc, Baltimore, Maryland, United States